CLINICAL TRIAL: NCT04140838
Title: Cost-utility and Physiological Effects of Acceptance and Commitment Therapy and Behavior Activation in Patients With Chronic Pain and Comorbid Major Depression (IMPACT Project)
Brief Title: Cost-utility and Physiological Effects of ACT and BATD in Patients With Chronic Pain and Depression
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Principal Investigator, Juan Vicente Luciano, Principal Investigator, Fundació Sant Joan de Déu
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI19/00112
Record Dates: First submitted 2019-10-22; First posted 2019-10-28 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Randomized Controlled Trial
MeSH Terms: interventions — Acceptance and Commitment Therapy; Therapeutics

STUDY DESIGN:
Intervention Model Description: Single-blind, parallel-group, randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TAU + Acceptance and Commitment Therapy (ACT) (Experimental): This therapy is based, as the name implies, on the acceptance (not avoidance) of negative experiences as a coping strategy, and on committing to life values or objectives. ACT has been used for various conditions, including chronic pain. Since avoidance is a strategy frequently used by patients suffering from pain, the application of this therapy seems very appropriate. In fact, it has been proven that patients who accept their pain more are those who score lower in pain intensity, have less negative emotions and enjoy a better quality of life.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT); Other: Treatment as Usual (TAU)
- TAU + Behavioral Activation Therapy for Depression (BATD) (Experimental): Behavioural and structured treatment based on the application of learning principles. Its objective is to counteract depressive symptoms and, as a consequence, to ensure that patients regain a productive and emotionally satisfying life. Its basic methodology consists in activating subjects with depression through programming and conduct of behaviours that are likely to increase the positive reinforcement of their context.
  Interventions: Behavioral: Behavioral Activation Therapy for Depression (BATD); Other: Treatment as Usual (TAU)
- Treatment as Usual (TAU) (Active Comparator): Standard Care. Although there is no treatment considered as the gold standard for chronic pain and comorbid major depression, the standard treatment is usually mainly pharmacological and conforms to the symptomatic profile of each patient.
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — Group treatment protocol of 8 weekly 90 minute sessions. Session 1: Presentation of the general concept of ACT therapy. Session 2: Value analysis I. Session 3: Value analysis II. Session 4: Value analysis III. Session 5: Values and feelings. Session 6: Taking a direction. Session 7: Dare and change. Session 8: Ready to act with ACT.
  Arms: TAU + Acceptance and Commitment Therapy (ACT)
Behavioral: Behavioral Activation Therapy for Depression (BATD) — Group treatment protocol of 8 weekly 90 minute sessions. Session 1: Collection of information regarding areas of activity and interaction contexts.
  Session 2: Identification of information related to depressive behaviours. Session 3 Obtaining complementary information regarding the characteristics of the history of patient interactions and any contexts.
  Session 4: Explanation of the hypotheses of problematic behaviour, its maintenance and change throughout the intervention.
  Session 5: Once the 10 target activities have been identified, a record is made to track and their progress weekly.
  Session 6: Discussion of what was obtained from the records in general and of the satisfaction obtained, and explanation of the contexts and reinforcers.
  Session 7: Psycho-education Session 8: New behaviours, the goals achieved and the maintenance of the weekly activity are inquired about.
  Arms: TAU + Behavioral Activation Therapy for Depression (BATD)
Other: Treatment as Usual (TAU) — Standard pharmacological treatment usually provided to patients suffering chronic pain and mild-moderate depression.

SUMMARY:
Objectives: (1) To analyze the effectiveness of adding a group-based form of Acceptance and Commitment Therapy (ACT) or a behavioural activation program for depression (TACD) to the treatment as usual (TAU) for patients diagnosed of chronic pain and comorbid mild-moderate major depression; (2) To examine the cost-utility of these psychological treatments from healthcare and societal perspectives; (3) To measure a set of biomarkers alongside the RCT in order to know the physiological underpinnings of these psychological therapies and to identify potential predictors of treatment response.

Methodology: 12-month multisite, randomised, controlled trial (RCT) Centres: Parc Sanitari Sant Joan de Déu (St. Boi de Llobregat) and Hospital del Mar (Barcelona).

Participants. 225 adult patients with chronic pain that meet the diagnostic criteria for mild-moderate major depression will be randomly assigned to one of the three study arms: TAU + ACT vs. TAU + TACD vs. TAU.

Primary outcome: Quality of life. Secondary outcomes: pain intensity, depression severity, anxiety symptoms, pain catastrophising, and pain acceptance. Costs to the healthcare system and to society and quality adjusted life years (QALYs). In addition, the empirically validated app Multicenter Pain Monitor® will be used to monitor participants alongside the treatments (ecological momentary assessment). Biomarkers: hair cortisol and cortisone, corticosteroid-binding globulin (CBG), ACTH and cortisol in plasma, and genotyping of 5 polymorphisms in the FKBP5 gene involved in the regulation of the hypothalamic-pituitary-adrenal axis activity, cytokines, Th1: IL-6, IL-8, TNF-α; cytokines Th2: IL-10 + hsCRP test, and vitamin D levels. Main statistical analyses: Intention-to-Treat analyses that will include all participants who undergo random allocation, using multiple imputation to replace missing values. Linear mixed-effects models will be performed using Restricted Maximum Likelihood to estimate the parameters. Calculation of between-groups effect sizes using Cohen's d and of the number-needed-to-treat. Economic evaluation: cost-utility ratios evaluated by applying bootstrapping techniques, acceptability curves, and sensitivity analyses.

DETAILED DESCRIPTION:
The IMPACT Project's main objective is to determine the effectiveness of adding to the standard care of patients with chronic pain and mild to moderate major depression a group programme based on ACT or a group programme based on BATD and analyse the cost-utility of these psychological treatments from a health and social perspective. Likewise, both in chronic pain and in other usually associated psychiatric diseases, there is a ubiquitous lack of knowledge about what specific psychological and physiological mechanisms are modified by these third generation psychotherapies and how they relate to the observed clinical results. The potential predictors of response to these treatments are also unknown. In chronic musculoskeletal pain where central sensitization plays an important role, alterations have been found in different markers associated with an increased experience of pain. Some of these alterations in markers (e.g. high levels of pro-inflammatory cytokines) would also appear to be shared with other psychiatric diseases (major depression), a fact that would suggest a possible common mechanism involved in the etiopathogenesis of these diseases. Third generation psychotherapies have proven effective for pain management and regulation of the immune response. The IMPACT Multicentre Project (Improving Pain and Depression with ACT and BATD) will significantly expand the limited knowledge available about how ACT and BATD therapies exert their effects on relevant clinical improvement variables and will try to identify response predictive factors to these treatments.

ELIGIBILITY:
Inclusion Criteria:

Patients who have been visited in the last 3 years in the participating centres and who have been given a diagnosis of chronic non-cancer musculoskeletal pain. In telephone screening, it will be evaluated whether the current pain intensity is at least moderate and PHQ-9 will be administered to confirm the presence of mild to moderate active depression.

1. Patients between 18 and 70 years of age.
2. Diagnosis of chronic pain (≥ 3 months) according to medical history (current pain ≥ 4 out of 10)
3. Diagnosis of mild to moderate depression according to PHQ-9 (score between 5 and 19).
4. Understanding of Spanish.
5. Access to a Smartphone (with Android operating system).
6. Written informed consent.

Exclusion Criteria:

1. Presence of cognitive impairment according to MMSE (≤ 24 out of 30).
2. Previous (last year) or current psychological treatment.
3. Presence of severe mental disorder (e.g. psychotic disorder) related to substance dependence/abuse or another disease that affects the CNS (organic brain pathology or head trauma of any severity).
4. Presence of serious, uncontrolled or degenerative medical disease that may interfere with affective symptoms.
5. Risk of suicide (Item 9 score of PHQ-9 ≥ 2).
6. Patients involved in legal proceedings with employers in relation to their illness.
7. Patients with scheduled surgical intervention or other interventions.
8. Inability to attend group treatment sessions.

Additional exclusion criteria for the study of biomarkers (50% of subjects in each branch):

1. Cold/infection symptoms on the day of blood collection.
2. Needle phobia.
3. BMI > 36 kg/m2 or weight > 110 kg
4. Consumption > 8 units of caffeine per day (maximum 1 drink with caffeine on the day of testing).
5. Smoker > 5 cigarettes a day.
6. Being pregnant or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Aggregate score of the Physical Function, Body Pain and Vitality subscales of the SF-36 | Through study completion, an average of 1 year
  The range of scores is 15 to 65. Higher scores indicate better quality of life.

SECONDARY OUTCOMES:
Numerical pain scale | Through study completion, an average of 1 year
  Patients evaluate their pain in a continuum from 0 to 10, where 0 is absence of pain and 0 is the worst possible pain.
Hospital Anxiety and Depression Scale (HADS) | Through study completion, an average of 1 year.
  Scale of 14 items created to assess symptoms of anxiety and depression. The total score ranges from 0 to 42, and each subscale (HADS-Anxiety and HADS-Depression) includes 7 items with scores ranging from 0 to 21. Higher scores indicate higher symptom severity.
Pain Catastrophising Scale (PCS) | Through study completion, an average of 1 year
  Scale of 13 items comprising three dimensions: rumination over pain, magnification of pain and helplessness in the face of pain symptoms. The PCS total score and subscale scores are computed as the sum of ratings for each item. This study used the total score, which can vary from 0 to 52 with higher scores indicating greater pain catastrophising.

OTHER OUTCOMES:
Psychological Inflexibility in Pain Scale (PIPS) | Through study completion, an average of 1 year
  12-item scale that assesses psychological inflexibility in patients with pain and includes two factors: avoidance and cognitive fusion with pain. For this study, only the total score is used; it ranges from 12 to 84, with higher scores indicating higher level of psychological inflexibility.
EuroQoL (EQ-5D-5L) | Through study completion, an average of 1 year
  Instrument for evaluating health-related quality of life. The EQ-5D-5L scores will be used to calculate the Quality-Adjusted Life Years (QALYs) for the cost-utility analysis
Behavioral Activation for Depression Scale (BADS) - short-form | Through study completion, an average of 1 year
  The BADS - short form consists of 9 items focusing on behavioral activation, each rated on a seven point scale ranging from 0 (not at all) to 6 (completely). Higher scores represent increased activation.
Credibility/Expectancy questionnaire (CEQ) | Baseline
  6-item questionnaire for measuring treatment expectancy and credibility for use in clinical outcome studies. Each item is rated from 0 to 10, with higher scores indicating better expectancy.
Client Service Receipt Inventory (CSRI) | Through study completion, an average of 1 year
  The version used in this study is designed to retrospectively collect information on the use of health and social services during the previous 12 months. This instrument does not provide total or sub-scale scores, only collects information about use of services and medication consumption.
Adverse effects of treatments | Through study completion, an average of 1 year
  Qualitative ad hoc measure to check the presence of negative effects of psychological treatments.
The Pain Monitor® app | Through study completion, an average of 1 year
  It has been recently validated in an empirical study for use on Android smartphones. It will be used to assess daily (twice a day) the level of pain, fatigue, catastrophism, etc. during the treatment period.
Socio-demographic questionnaire | Baseline
  Gender, date of birth, marital status, living arrangements, educational level and employment status.
Patient Health Questionnaire (PHQ-9) | Baseline
  PRIME-MD module with 9 items adjusted to the DSM-IV criteria for major depression. It can be used algorithmically for the probable diagnosis of a depressive disorder, or as a continuous measure of scores ranging from 0 to 27, with cut-off points of 5, 10, 15 and 20, which set the levels of symptoms of depression as mild, moderate, moderately severe or severe.

CONTACTS AND LOCATIONS:
Overall Officials: Juan V. Luciano, PhD, Principal Investigator — Fundació Sant Joan de Déu
Locations (2):
- Spain (2):
  - Parc Sanitari Sant Joan de Déu (PSSJD), Sant Boi de Llobregat, Barcelona
  - Parc de Salut Mar, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanabria-Mazo JP, Forero CG, Cristobal-Narvaez P, Suso-Ribera C, Garcia-Palacios A, Colomer-Carbonell A, Perez-Aranda A, Andres-Rodriguez L, McCracken LM, D'Amico F, Estivill-Rodriguez P, Carreras-Marcos B, Montes-Perez A, Comps-Vicente O, Esteve M, Grasa M, Rosa A, Cuesta-Vargas AI, Maes M, Borras X, Edo S, Sanz A, Feliu-Soler A, Castano-Asins JR, Luciano JV. Efficacy, cost-utility and physiological effects of Acceptance and Commitment Therapy (ACT) and Behavioural Activation Treatment for Depression (BATD) in patients with chronic low back pain and depression: study protocol of a randomised, controlled trial including mobile-technology-based ecological momentary assessment (IMPACT study). BMJ Open. 2020 Jul 23;10(7):e038107. doi: 10.1136/bmjopen-2020-038107. PMID 32709656
- [Result] Sanabria-Mazo JP, Colomer-Carbonell A, Borras X, Castano-Asins JR, McCracken LM, Montero-Marin J, Perez-Aranda A, Edo S, Sanz A, Feliu-Soler A, Luciano JV. Efficacy of Videoconference Group Acceptance and Commitment Therapy (ACT) and Behavioral Activation Therapy for Depression (BATD) for Chronic Low Back Pain (CLBP) Plus Comorbid Depressive Symptoms: A Randomized Controlled Trial (IMPACT Study). J Pain. 2023 Aug;24(8):1522-1540. doi: 10.1016/j.jpain.2023.04.008. Epub 2023 Apr 25. PMID 37105508
- [Derived] Sanabria-Mazo JP, D'Amico F, Cardenosa E, Ferrer M, Edo S, Borras X, McCracken LM, Feliu-Soler A, Sanz A, Luciano JV. Economic Evaluation of Videoconference Group Acceptance and Commitment Therapy and Behavioral Activation Therapy for Depression Versus Usual Care Among Adults With Chronic Low Back Pain Plus Comorbid Depressive Symptoms. J Pain. 2024 Jul;25(7):104472. doi: 10.1016/j.jpain.2024.01.337. Epub 2024 Jan 18. PMID 38242333